CLINICAL TRIAL: NCT02159586
Title: Cardiac Vagal Effects of Gastric Electrical Stimulation and Vagal Nerve Action Potentials in Vagus Nerve in Patients With Gastroparesis
Brief Title: Cardiac Vagal Effects of GES in Patients With Gastroparesis and Vagal Nerve Action Potentials in Vagus Nerve
Acronym: GES
Status: Active, not recruiting | Type: Observational
Sponsor: Indiana University (Other)
Collaborators: Purdue University (Other)
Responsible Party: Principal Investigator, Thomas V. Nowak, MD, Indiana University
Other Study IDs: EKG/Vagal Nerve; 1206008988 (Other: IRB)
Record Dates: First submitted 2014-06-06; First posted 2014-06-10 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Gastroparesis
Keywords: gastroparesis; gastric electrical stimulator; GES; vomiting; nausea; bloating; postprandial fullness; epigastric pain
MeSH Terms: conditions — Gastroparesis; Vomiting; Nausea

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Blood will be withdrawn to assess the hormones like insulin, cholecystokinin and serotonin
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- GES subjects: male and female patients at least 18 years of age, with gastroparesis, who will or have already undergone the implantation of a GES device
  Interventions: Device: gastric electrical stimulator

INTERVENTIONS:
Device: gastric electrical stimulator

SUMMARY:
The objective of this study is to determine if Gastric Electrical Stimulation may influence vagal outflow via vagal afferent fibers that terminate in the Central Nervous System.

DETAILED DESCRIPTION:
All patients who are going to have a GES device implanted, or who already have the device are eligible to be part of the study. They will be followed according to the time point they enter the study and its schedule. The visit procedures will be conducted at the discretion of the investigator dependent on the clinical condition of the subject at that time. The study involves EKG and vagal nerve recordings. Three EKG electrodes will be placed (one on chest and 2 on either arms or legs). Separate electrodes will be placed on the neck overlying the vagus nerves

Baseline Visit:

Subjects who are being seen in clinic for possible gastroparesis and may be a possible candidate for GES later or will be undergoing the GES implantation may have a baseline visit. . The baseline visit can be held either at the time of the clinic visit or before the GES implantation. If the baseline visit occurs on the day of the GES implantation, 2 separate EKGs will be performed, one prior to GES pacemaker device implantation for upto a duration of 5 minutes and the second one after the implantation in the recovery room. This EKG will be performed for a total duration of upto 15 minutes with 5 minute "ON", 5 minutes :OFF" and another 5 minutes in the "ON" position. At the same visit with each EKG recording separate EKG electrode will be placed on the neck overlying the vagus nerve. Vagal nerve recordings will be documented for a total duration of upto 15 minutes with approximately 5 min at "ON", 5 min "OFF" and another 5 min "ON" settings of the stimulator in conjunction with the EKG recordings.

At the baseline visit separate EKG electrodes will also be placed on the neck overlying the vagus nerve and a 5 minute recording will be made in conjunction with the EKG recordings.\ before the implantation.

If the subjects already have the GES device implanted then a baseline visit will not be required. They will be included in the study at the time the consent form is signed and will be followed as needed according to the clinic visit schedule and at the discretion and clinical judgement of the investigator

Post-implant Visits:

The subject may be asked at the clinic visits to repeat the EKG and vagal nerve study procedures at the discretion and clinical judgment of the investigator.

Identified patients will be contacted by the research team before their scheduled clinic visit and given the information about the study. If they agree verbally to participate then they will be asked to not have anything to eat or drink past 10pm the night before the appointment. They can take some water and medications as needed. The patients will physically sign the consent document on the day of the visit before the start of any procedures.

At the post GES pacemaker device implantation visit electrocardiogram (EKG) and the vagal nerve recording may be conducted.

Identified patients will be contacted by the research team before their scheduled clinic visit and given the information about the study. If they agree verbally to participate, then they will be asked to not have anything to eat or drink past 10 pm the night before the appointment. They can take some water and medications as needed. The patients will physically sign the consent document on the day of the visit before the start of any procedures.

EKG electrodes will be placed on the chest and arms/legs, and vagal nerve electrodes will be placed on the neck overlying the vagus nerve. A butterfly catheter is inserted under aseptic conditions into a peripheral vein. Fifteen ml (1 tablespoon) of blood is withdrawn and placed on ice (labeled Baseline). With the subject at rest recordings may be made for upto a total duration of 15- 20 minutes. After 15- 20 minutes of recordings the GES device is then turned "OFF" and recordings will be made for up to 40 minutes. After 40 minutes additional 15 ml (1 tablespoon) of blood is withdrawn after the device has been in the OFF position for 40 minutes (labeled "OFF"). The device is then turned back in the "ON" position with the GES settings either at the original or changed settings from the previous settings based on the clinical judgement of the investigators, The EKG and vagal recordings may be made for up to 15-20 minutes. After 15- 20 minutes in the ON position 15 ml (1 tablespoon) is then withdrawn (labeled "ON". The butterfly catheter is then withdrawn, and a bandage is placed at the venipuncture site. The final setting on the GES will depend on the clinical decision of the investigator based on the subject's symptoms and presentation to the clinic.

Another part of the study is to determine the best method and place for the placement of the electrodes on the neck overlying the vagus nerve. For this either an ultrasound machine (an imaging method that uses sound waves to create pictures of the inside of your body) or a digital stethoscope ( a device that is used to listen to your heart by your physician) will be used to find the carotid artery on the side of the neck. The vagus nerve lies approximately over or to the side of the carotid artery and the ultrasound machine will thus be able to help us identify the approximate place where the vagus nerve is close to the skin in the neck.

Subjects may be asked to undergo an ultrasound of the neck region or have a digital stethoscope placed over the neck to find the exact location of the carotid artery and thus the vagus nerve before the electrodes are placed. First, a tape measure will be used to measure neck circumference and neck length. The tape will be placed around the neck above the Adam's apple (region in front of the neck that feels bony and is more prominent in men than women) to measure the circumference. To measure neck length the tape will be placed from below the chin to the top of the chest. The subjects neck will be palpated to locate the proper landmarks.

The electrodes on the subjects neck will be placed according to the traditional method by feeling for the carotid artery and a 5 minute recording will be made.

After this the ultrasound machine will be used to find the carotid artery and hence the vagus nerve. The electrodes will then be placed according to the information from the ultrasound machine and another 5 minute of recording will be made.

To find the carotid artery using the stethoscope/ ultrasound, machine will be moved at several places on the neck and the place where the device shows the highest measurement will be used as the point where the carotid artery or the vagus nerve is most superficial. You may be asked to move your neck to one side or raise your chin up to find the best location.

If the subjects are taking part in the ultrasound guided / stethoscope method of electrode placement, then they will not be required to complete the other parts of the study.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Documented diagnosis of gastroparesis.
* Will undergo implantation of a GES device or already has a GES device implanted

Exclusion Criteria:

* Pregnancy
* History of allergic reaction to EKG lead placement adhesives.
* unable to give informed consent

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will evaluate male and female patients at least 18 years of age, with gastroparesis, who will or have already undergone the implantation of a GES device (Enterra, Medtronic, Minneapolis, MN)
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2012-11; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determine if GES influences vagal outflow | 2-3 years
  To determine if GES may influence vagal outflow via vagal afferent fibers that terminate in the Central Nervous System; EKG electrodes will be placed on the chest, stomach, jugular, and vagas nerves. The purpose of this is to record the effects of the stimulator when on and off. The ECG signals are digitized with an ECG power amplifier, Power Lab by AD Instruments. The digitized signals are analyzed with an ECG software analysis system, Lab Chart. The analysis will look for heart rate variability, total power variability, and frequency variability. This will determine if stimulation has an effect on these levels.

SECONDARY OUTCOMES:
Release of hormones | 2-3 years
  The purpose of this investigation is to determine whether gastric electrical stimulation of the stomach via a surgically implanted stimulation device is associated with gastrointestinal hormone release in human subjects. Blood draws will be obtained in tandem with each of the 3 phases of EKG recordings. The blood samples will be processed and serum will be sent to an IU Lab for Hormone analysis to see if typical hormone levels associated with digestion increase or decrease with the addition/subtraction of the gastric stimulation.
Vagus nerve anatomy | 2-3 years
  To optimize the methods for determining electrode placement around the cervical vagus nerve. The development of a method to record and analyze compound action potentials from the vagus nerve will enhance our knowledge of the mechanism of action of VNS in the treatment of gastroparesis.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Nowak, MD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No